CLINICAL TRIAL: NCT05026866
Title: A Study of Donanemab Versus Placebo in Participants at Risk for Cognitive and Functional Decline of Alzheimer's Disease
Brief Title: A Donanemab (LY3002813) Study in Participants With Preclinical Alzheimer's Disease (TRAILBLAZER-ALZ 3)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18284; I5T-MC-AACM (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — donanemab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donanemab (Experimental): Donanemab administered intravenously (IV)
  Interventions: Drug: Donanemab
- Placebo (Placebo Comparator): Placebo is administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donanemab — Administered intravenously
  Other Names: LY3002813
  Arms: Donanemab
Drug: Placebo — Administered intravenously
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of donanemab in participants with preclinical Alzheimer's Disease (AD) over up to 332 weeks. Approximately 800 additional participants will be enrolled in the 12-month Addendum 7 to assess safety of a different titration regimen.

ELIGIBILITY:
Inclusion Criteria:

* A Telephone Interview for Cognitive Status - modified (TICS-M) score reflective of intact cognitive functioning.
* Has a phosphorylated tau (P-tau) result consistent with the presence of amyloid pathology.
* Has a reliable study partner and backup study partner familiar with overall function and behavior, such as day-to-day activities and cognitive abilities.
* Have adequate literacy, vision, and hearing for neuropsychological testing at screening.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Female participants include those who are infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as Mullerian agenesis; or post menopausal (women 55 or older not on hormone therapy and had at least 12 months of spontaneous amenorrhea; or with a diagnosis of menopause prior to starting hormone replacement therapy.

Treatment Extension: (Study Period II Placebo Group Only)

* Are actively participating in Study AACM at the conclusion of Study Period III.

Exclusion Criteria:

* Mild cognitive impairment or dementia, or significant other neurodegenerative disease that can affect cognition.
* Current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, psychiatric, immunologic, or hematologic disease that could interfere with the analysis of the study or a life expectancy of approximately ≤5 years.
* History of cancer with high risk of recurrence and preventing completion of the trial.
* History of clinically significant multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions (including but not limited to erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and/or exfoliative dermatitis).
* Have any clinically important abnormality at screening on magnetic resonance imaging (MRI) or clinical laboratory test results that could be detrimental to the participant or study integrity.
* Have any contraindications for MRI, including claustrophobia or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemaker.
* Have a centrally read MRI demonstrating presence of amyloid-related imaging abnormalities (ARIA-E), >4 cerebral microhemorrhages, more than 1 area of superficial siderosis, any macrohemorrhage or severe white matter disease at screening.
* Have had prior treatment with a passive anti-amyloid immunotherapy <5 half-lives prior to randomization.
* Have received active immunization against amyloid beta (Aβ) in any other study.
* Have received active immunization against Aβ in any other study.
* Current or previous use of prescription medications used as treatment for mild cognitive impairment (MCI) or AD.

Addendum 7 Exclusion Criteria:

* Same as the main study except contraindications for florbetapir F 18 PET are exclusionary.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2996 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Progression of Composite Endpoint as Measured by Clinical Dementia Rating (CDR) in the Primary Study Population (Baseline CDR-Global Score [GS 0]) | Estimated up to Week 332
  Time to clinical progression as measured by CDR. CDR is a clinician-rated scale that provides an overall assessment of the participant's stage on the spectrum of Alzheimer's Disease (AD) dementia

SECONDARY OUTCOMES:
Change from Baseline in Cognitive Composite in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in Cognitive Composite in the Primary Study Population (CDR-GS 0)
Change from Baseline in International Shopping List Test (ISLT) in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in clinical progression as measured by ISLT in the Primary Study Population (Baseline CDR-GS 0)
Change from Baseline in Continuous Paired Associate Learning (CPAL ) in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in clinical progression as measured by CPAL in the Primary Study Population (baseline CDR-GS 0)
Change from Baseline in International Daily Symbol Substitution Test-Medicines (iDSSTm) in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in clinical progression as measured by iDSSTm in the Primary Study Population (Baseline CDR-GS 0)
Change from Baseline in Category Fluency in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in clinical progression as measured by Category Fluency in the Primary Study Population (Baseline CDR-GS 0)
Change from Baseline in CDR-Sum of Boxes (CDR-SB) n the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up Week 332
  Change from baseline in clinical progression as measured by CDR-SB in the Primary Study Population (Baseline CDR-GS 0)
Change from Baseline in Cognitive Function Index (CFI) in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in clinical progression as measured by CFI in the Primary Study Population (Baseline CDR-GS 0)
Change from Baseline in Montreal Cognitive Assessment (MoCA) Score in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in clinical progression as measured by MoCA score in the Primary Study Population (Baseline CDR-GS 0)
Change from Baseline in Mild Behavioral Impairment Checklist (MBI-C) in the Primary Study Population (Baseline CDR-GS 0) | Baseline, Up to Week 332
  Change from baseline in MBI-C in the Primary Study Population (Baseline CDR-GS 0)
Time to Clinical Progression of Composite Endpoint as Measured by CDR in the Overall Study Population (Baseline CDR-GS 0 or 0.5) | Baseline, Up to Week 332
  Time to clinical progression as measured by CDR in the Overall Study Population (Baseline CDR-GS 0 or 0.5)
Time to Clinical Progression as Measured by CDR Memory Box in Primary Study Population (Baseline CDR-GS 0) | Estimated up to Week 332
  Time to clinical progression as measured by CDR Memory Box in the Primary Study Population (Baseline CDR-GS 0)
Time to Clinical Progression as Measured by CDR Judgment and Problem Solving Box in the Primary Study Population (Baseline CDR-GS 0) | Estimated up to Week 332
  Time to clinical progression as measured by CDR Judgment and Problem Solving Box in the Primary Study Population (Baseline CDR-GS 0)
Time to Clinical Progression as Measured by At Least 0.5 Change on CDR-SB in Primary Study Population (Baseline CDR-GS 0) | Estimated up to Week 332
  Time to clinical progression as measured by at least 0.5 change on CDR-SB in Primary Study Population (Baseline CDR-GS 0)
Time to Clinical Progression of Composite Endpoint as Measured by CDR in Subpopulation Positive Based on Secondary Diagnostic Test | Estimated up to Week 332
  Time to clinical progression as measured by CDR in subpopulation positive based on secondary diagnostic test
Change from Baseline in Plasma P-tau217 | Baseline, Up to Week 332
  Change from baseline in Plasma P-tau217
Pharmacokinetics (PK): Average Serum Donanemab Concentration at Steady State | Baseline through Week 76
  PK: Average serum donanemab concentration at steady state
Percentage of Participants with Treatment-emergent Anti-Drug Antibody (ADAs) | Baseline through Week 16
  Percentage of participants with treatment-emergent anti-drug antibody (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (216):
- United States (198):
  - Parkway Medical Center, Birmingham, Alabama
  - Alabama Psychiatry - Birmingham - Brookwood Medical Center Drive, Homewood, Alabama
  - Rehabilitation & Neurological Services, Huntsville, Alabama
  - Care Access - 801 South Power Road, Mesa, Mesa, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Alzheimer's Institute Tucson, Tucson, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Care Access - Berkeley, Berkeley, California
  - Care Access - Beverly Hills, Beverly Hills, California
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - Valley Clinical Trials, Inc., Covina, California
  - Neurology Center of North Orange County, Fullerton, California
  - Care Access - Gilroy, Gilroy, California
  - Marvel Clinical Research, Huntington Beach, California
  - Care Access Research - Huntington Beach, Huntington Beach, California
  - Irvine Clinical Research, Irvine, California
  - Option Care - Irvine, Irvine, California
  - Kaizen Brain Center, La Jolla, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Pacific Research Network, Lemon Grove, California
  - Healthy Brain Clinic, Long Beach, California
  - Neurovations, Napa, California
  - Care Access - Newport Beach, Newport Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Inland Psychiatric Medical Group, Redlands, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Option Care - Riverside, Riverside, California
  - Clinical Trials Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Ray Dolby Brain Health Center, San Francisco, California
  - Care Access - Los Gatos, San Jose, California
  - Syrentis Clinical Research, Santa Ana, California
  - Care Access - Santa Clarita, Santa Clarita, California
  - Option Care - Los Angeles South, Santa Fe Springs, California
  - Providence Medical Foundation, Santa Rosa, California
  - Mazur, Statner, Dutta, Nathan, PC, Thousand Oaks, California
  - Tilda Research, Tustin, California
  - Velocity Clinical Research, Panorama City, Van Nuys, California
  - Infectious Disease Doctors Medical Group, APC, Walnut Creek, California
  - Care Access - Aurora, Aurora, Colorado
  - Mountain Neurological Research Center, Basalt, Colorado
  - Denver Neurological Research, Denver, Colorado
  - Invicro, New Haven, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - SFM Clinical Research, Boca Raton, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Care Access - Daytona Beach, Daytona Beach, Florida
  - Care Access - Delray Beach, Delray Beach, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Care Access - Guava Street, Lady Lake, Florida
  - Accel Research Sites - St. Pete-Largo Clinical Research Unit, Largo, Florida
  - ClinCloud - Maitland, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - ClinCloud - Viera, Melbourne, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Optimus U Corporation, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - VIN-Andrew Lerman, Miami, Florida
  - South Florida Research Phase I-IV, Miami, Florida
  - Brainstorm Research Group, Miami, Florida
  - IMIC, Inc., Miami, Florida
  - VIN-Victor Faradji, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - VIN- Margarita Almeida El-Ramey, Pembroke Pines, Florida
  - Emerald Coast Neurology - Airport Boulevard, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Care Access - Tamarac, Tamarac, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Vicis Clinical Research, Tampa, Florida
  - Care Access - Tampa, Tampa, Florida
  - Coram CVS/Specialty Infusion Services - Tampa, Tampa, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Masters of Clinical Research, Augusta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - SKY Clinical Research Network Group-Blake, Union City, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - IMA Clinical Research Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - AMITA Health - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Care Access - Fairview Heights, Fairview Heights, Illinois
  - Great Lakes Clinical Trials - Gurnee, Gurnee, Illinois
  - Accellacare - DuPage, Lombard, Illinois
  - Coram CVS/Specialty Infusion Services - Fort Wayne, Fort Wayne, Indiana
  - Care Access - South Indianapolis, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Covenant Medical Center, Waterloo, Iowa
  - College Park Specialty Center, Overland Park, Kansas
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Optum Infusion - Baton Rouge, Baton Rouge, Louisiana
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Care Access - Quincy, Quincy, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Revival Research Institute, Southfield, Michigan
  - Minneapolis Clinic of Neurology - Burnsville Office, Burnsville, Minnesota
  - Coram CVS/Specialty Infusion Services - Mendota Heights, Mendota Heights, Minnesota
  - SKY Clinical Research Network Group - Hall, Fayette, Mississippi
  - SKY Clinical Research Network Group-Quinn, Ridgeland, Mississippi
  - Citizens Memorial Hospital District, Bolivar, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - IMA Clinical Research - St. Louis, St Louis, Missouri
  - Coram CVS/Specialty Infusion Services - Henderson, Henderson, Nevada
  - Option Care - Las Vegas, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - IMA Clinical Research Hoboken, Hoboken, New Jersey
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - IMA Clinical Research Albany, Albany, New York
  - Neurological Associates Albany, Albany, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - IMA Clinical Research Westchester, Hartsdale, New York
  - IMA Clinical Research, New York, New York
  - South Shore Neurologic Associates, Patchogue, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Prime Global Research, The Bronx, New York
  - Asheville Neurology Specialists, Asheville, North Carolina
  - Care Access - Charlotte, Charlotte, North Carolina
  - Care Access - Fayetteville, Fayetteville, North Carolina
  - Care Access - Greensboro, Greensboro, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Care Access - Kinston, Kinston, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Care Access - Raleigh, Raleigh, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - Hometown Urgent Care and Research - Cincinnati, Dayton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Care Access - Lima, Lima, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Care Access - Youngstown, Poland, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Optum Infusion - Bend, Bend, Oregon
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Center for Cognitive Health, Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Care Access - Pottsville, Pottsville, Pennsylvania
  - Care Access Research - Warwick, Warwick, Rhode Island
  - Care Access - Anderson, Anderson, South Carolina
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - VitaLink Research - Columbia, Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - VitaLink Research - Greenville, Greenville, South Carolina
  - Care Access - Mauldin, Mauldin, South Carolina
  - VitaLink Research - Spartanburg, Spartanburg, South Carolina
  - VitaLink Research - Union, Union, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Neurology Clinic, Cordova, Tennessee
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Memphis, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Senior Adults Specialty Research, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Headlands Research - Brownsville, Brownsville, Texas
  - Conroe Willis Medical Research, Conroe, Texas
  - Advanced Neuro Research Center - ANRC, El Paso, Texas
  - Care Access - Georgetown, Georgetown, Texas
  - Optum Infusion - Houston, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - Family Practice Center, McAllen, Texas
  - El Faro Health and Therapeutics, Rio Grande City, Texas
  - Benchmark Research - Knickerbocker, San Angelo, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - The Memory Clinic, Bennington, Vermont
  - Care Access - Arlington, Arlington, Virginia
  - Option Care - Chantilly, Chantilly, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Universal Research Group, Tacoma, Washington
  - Optum Infusion - Woodinville, Woodinville, Washington
  - Exemplar Research, Morgantown, West Virginia
- Japan (12):
  - The University of Tokyo Hospital, Bunkyō City
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Tokyo Asbo Clinic, Chūōku
  - P-One Clinic, Hachiōji
  - AMC Nishiumeda Clinic, Osaka
  - National Center for Geriatrics and Gerontology, Ōbu
  - Samoncho Clinic, Shinjuku
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi
  - Tokyo Metropolitan Geriatric Hospital, tabashi City
  - Oita University Hospital, Yufu
- Puerto Rico (6):
  - SCB Research Center, Bayamón
  - Dr. Samuel Sanchez PSC, Caguas
  - INSPIRA Clinical Research, San Juan
  - Instituto De Neurologia Dra. Ivonne Fraga, San Juan
  - Mindful Medical Research, San Juan
  - University of Puerto Rico - Medical Sciences Campus_Do not use - Duplicate facility, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Yaari R, Holdridge KC, Williamson M, Wessels AM, Shcherbinin S, Kotari V, Reiman EM, Tariot PN, Alexander R, Langbaum JB, Sims JR. Donanemab in preclinical Alzheimer's disease: Screening and baseline data from TRAILBLAZER-ALZ 3. Alzheimers Dement. 2025 Sep;21(9):e70662. doi: 10.1002/alz.70662. PMID 40955720
- See also: A Donanemab (LY3002813) Prevention Study in Participants With Alzheimer's Disease (TRAILBLAZER-ALZ 3) — https://trials.lillytrialguide.com/en-US/trial/vpJyQXuNAxTOFoL7o2Gbk